CLINICAL TRIAL: NCT07301086
Title: Deep Learning-Assisted Ultrasonic Diagnosis and Localization of Testicular Appendix Torsion: A Multicenter Retrospective Validation Study
Brief Title: Deep Learning-Assisted Ultrasonic Diagnosis and Localization of Testicular Appendix Torsion
Status: Not yet recruiting | Type: Observational
Sponsor: Ying Jiang (Other)
Responsible Party: Sponsor-Investigator, Ying Jiang, resident physician, The Children's Hospital of Zhejiang University School of Medicine
Organization: The Children's Hospital of Zhejiang University School of Medicine (Other)
Other Study IDs: CHZhejiangjiangying
Record Dates: First submitted 2025-12-09; First posted 2025-12-24 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Testicular Appendix Torsion; Testicular Torsion; Epididymitis
Keywords: Testicular Appendix Torsion; Deep Learning; Ultrasonic Diagnosis
MeSH Terms: conditions — Spermatic Cord Torsion; Epididymitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Testicular Appendix Torsion Group: Patients diagnosed with testicular appendage torsion
- Testicular Torsion Group: Patients diagnosed with testicular torsion
- Epididymitis Group: Patients diagnosed with epididymitis
- Normal Group: Patients with no testicular appendage torsion,testicular torsion,epididymitis,and the scrotum is normal

SUMMARY:
Ultrasound data were both retrospectively and prospectively collected from the primary center and six other sub-centers. Combined with clinical diagnostic outcomes, the data labeling was completed by physicians with extensive clinical experience. In this study, ConvNeXtV2 was used as the classification network and YOLOv12 was adopted as the detection network.The retrospective dataset from the primary center was split into training, validation, and test subsets, on which the model was trained, validated, and tested respectively; additional validation was conducted on both retrospective and prospective datasets from the primary center and sub-centers.Meanwhile, four physicians were assigned to interpret the ultrasound data from the retrospective and prospective datasets from the primary center and sub-centers using two diagnostic methods-independent diagnosis and artificial intelligence (AI)-assisted diagnosis-and the diagnostic accuracy of these two approaches was further compared.By collecting and learning the treatment methods of patients in the primary center training set, predicting the treatment methods of patients in the sub-center datasets, and comparing the proportion of surgeries predicted by AI with the actual proportion of surgeries, the efficacy of the model was verified.

DETAILED DESCRIPTION:
Ultrasound data were both retrospectively and prospectively collected from the primary center and six other sub-centers. Combined with clinical diagnostic outcomes, the data labeling was completed by physicians with extensive clinical experience. In this study, ConvNeXtV2 was used as the classification network and YOLOv12 was adopted as the detection network.The retrospective dataset from the primary center was split into training, validation, and test subsets, on which the model was trained, validated, and tested respectively; additional validation was conducted on both retrospective and prospective datasets from the primary center and sub-centers.Meanwhile, four physicians were assigned to interpret the ultrasound data from the retrospective and prospective datasets from the primary center and sub-centers using two diagnostic methods-independent diagnosis and artificial intelligence (AI)-assisted diagnosis-and the diagnostic accuracy of these two approaches was further compared.By collecting and learning the treatment methods of patients in the primary center training set, predicting the treatment methods of patients in the sub-center datasets, and comparing the proportion of surgeries predicted by AI with the actual proportion of surgeries, the efficacy of the model was verified.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 18 years old
2. Underwent ultrasound examination due to acute scrotal pain (≤ 24 hours)
3. Patients clinically diagnosed with testicular appendage torsion (TAT)

Exclusion Criteria:

1. Poor ultrasound image quality (failure to identify testicular structures)
2. Incomplete clinical data (failure to confirm the diagnosis of testicular appendage torsion [TAT])

Ages: 1 Minute to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Biological male
Study Population: Age ≤ 18 years old，underwent ultrasound examination due to acute scrotal pain (≤ 24 hours)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of deep-learning model verify four conditions:testicular appendage torsion;testicular torsion;epididymitis and normal condition | From image input to result generation is expected to be 24 hours
  accuracy of deep-learning model verify four conditions:testicular appendage torsion;testicular torsion;epididymitis and normal condition

SECONDARY OUTCOMES:
Number of Participants with Acute Scrotal Pain | From enrollment begin to the end is expected to be 5 months
The accuracy rate of clinicians in diagnosing and localizing testicular appendix torsion | From the begin of Clinicians diagnose and locate to the end is expected to be 15 days
The accuracy rate of the Deep learning model in predicting the treatment modality for testicular appendix torsion,conservative treatment or surgery | From the begin of the prediction of treatment for testicular appendix torsion by Deep learning model to the end is expected to be 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing Ye, Phd Degree, Study Director — Zhejiang University School of Medicine Children's Hospital
Locations (1):
- Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
the patient's ultrasound images and baseline data
Supporting Information: Study Protocol
Time Frame: The IPD and supporting information will be available at 1st Jan,2027, and for one month
Access Criteria: Journal editors and reviewers,study protocol,send me email to access it.